CLINICAL TRIAL: NCT01895335
Title: A Prospective, Single-Arm, Clinical-Setting Study to Describe Efficacy, Tolerability and Convenience of Teriflunomide Treatment Using Patient Reported Outcomes (PROs) in Relapsing Multiple Sclerosis (RMS) Patients
Brief Title: Using Patient Reported Outcomes (PROs) to Evaluate Teriflunomide Treatment in Relapsing Multiple Sclerosis (RMS) Patients
Acronym: TERI-PRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS13567; U1111-1139-8730 (Other: UTN)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teriflunomide (Experimental): Teriflunomide 14 mg or 7 mg according to local labelling once daily (QD) orally for 48 weeks.
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — Pharmaceutical form: film-coated tablet; Route of administration: oral
  Other Names: HMR1726; Aubagio®

SUMMARY:
Primary Objective:

To describe efficacy, tolerability and convenience of teriflunomide treatment through the evaluation of Participant Reported Outcomes (PROs).

Secondary Objectives:

To describe disease progression using PROs. To describe clinical outcomes (ie, treated relapses) in teriflunomide treated participant.

To describe the change in cognition in teriflunomide treated participants. To describe safety of teriflunomide in participant treated (based on adverse events reporting).

To describe adherence and persistence to teriflunomide treatment. To describe quality of life, activity and leisure over the period of teriflunomide treatment.

To compare Participant Determined Disease Steps (PDDS) and Expanded Disability Status Scale (EDSS) in assessing Multiple Sclerosis (MS) disease progression.

DETAILED DESCRIPTION:
The total duration of the study per participant was up to 50 or 54 weeks (if accelerated elimination procedure performed):

Screening: up to 2 weeks Teriflunomide treatment: 48 weeks Accelerated elimination procedure: 4 weeks when performed

An accelerated elimination procedure at any time after discontinuation of teriflunomide treatment was possible and it was particularly recommended for women of child-bearing potential.

ELIGIBILITY:
Inclusion criteria:

Participants with a relapsing form of multiple sclerosis (RMS) having signed written informed consent.

Exclusion criteria:

* According to local labelling,
* Less than 18 years of age,
* Current or history of receiving teriflunomide,
* Previous treatment with leflunomide within 6 months prior to baseline,
* Participants with preexisting acute or chronic liver disease, or those with serum alanine aminotransferase (ALT) greater than 2 times the upper limit of normal (ULN),
* Known history of active tuberculosis (TB) or latent TB infection, either diagnosed by standard medical practice or guidelines (including skin or blood test, chest X-ray, or as appropriate per local practice),
* Known history of severe immunodeficiency, acquired immunodeficiency syndrome (AIDS), bone marrow disease, acute or severe active infections,
* Women who were pregnant or breast-feeding,
* Female participants with a positive pregnancy test at screening or women of child-bearing potential who did not agree to use reliable contraception throughout the course of the study,
* Male participants (only when required according to local labeling): unwilling to use reliable contraception during the course of the study,
* Additional exclusion criteria applicable for Europe (EU) countries (in accordance with contraindications of EU summary of product characteristics [SmPC]):

  * Participants with significantly impaired bone marrow function or significant anaemia, leukopenia, neutropenia or thrombocytopenia,
  * Participants with severe active infection until resolution,
  * Participants with severe renal impairment undergoing dialysis, because insufficient clinical experience was available in this participant group,
  * Participants with severe hypoproteinaemia, e.g. in nephrotic syndrome.
* Hypersensitivity to the active substance or to any of the excipients,
* Other additional contraindications per local labeling.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (169):
- United States (75):
  - Investigational Site Number 840077, Birmingham, Alabama
  - Investigational Site Number 840007, Cullman, Alabama
  - Investigational Site Number 840087, Phoenix, Arizona
  - Investigational Site Number 840114, Phoenix, Arizona
  - Investigational Site Number 840080, Scottsdale, Arizona
  - Investigational Site Number 840032, Tucson, Arizona
  - Investigational Site Number 840021, Phoenix, Arkansas
  - Investigational Site Number 840018, Fullerton, California
  - Investigational Site Number 840037, Fullerton, California
  - Investigational Site Number 840108, Long Beach, California
  - Investigational Site Number 840014, Newport Beach, California
  - Investigational Site Number 840019, Oceanside, California
  - Investigational Site Number 840097, Boulder, Colorado
  - Investigational Site Number 840040, Colorado Springs, Colorado
  - Investigational Site Number 840046, Denver, Colorado
  - Investigational Site Number 840016, Englewood, Colorado
  - Investigational Site Number 840094, Fort Collins, Colorado
  - Investigational Site Number 840024, Bradenton, Florida
  - Investigational Site Number 840089, Clearwater, Florida
  - Investigational Site Number 840055, Coconut Creek, Florida
  - Investigational Site Number 840104, Hialeah, Florida
  - Investigational Site Number 840101, Miami Lakes, Florida
  - Investigational Site Number 840011, Ormond Beach, Florida
  - Investigational Site Number 840059, Sarasota, Florida
  - Investigational Site Number 840008, St. Petersburg, Florida
  - Investigational Site Number 840081, Sunrise, Florida
  - Investigational Site Number 840002, Atlanta, Georgia
  - Investigational Site Number 840075, Macon, Georgia
  - Investigational Site Number 840012, Fort Wayne, Indiana
  - Investigational Site Number 840010, Indianapolis, Indiana
  - Investigational Site Number 840034, Louisville, Kentucky
  - Investigational Site Number 840047, Rockport, Maine
  - Investigational Site Number 840107, Foxborough, Massachusetts
  - Investigational Site Number 840030, Springfield, Massachusetts
  - Investigational Site Number 840073, Clinton Township, Michigan
  - Investigational Site Number 840068, Golden Valley, Minnesota
  - Investigational Site Number 840098, Golden Valley, Minnesota
  - Investigational Site Number 840086, Chesterfield, Missouri
  - Investigational Site Number 840058, St Louis, Missouri
  - Investigational Site Number 840026, Lincoln, Nebraska
  - Investigational Site Number 840020, Henderson, Nevada
  - Investigational Site Number 840049, Freehold, New Jersey
  - Investigational Site Number 840044, Toms River, New Jersey
  - Investigational Site Number 840100, East Setauket, New York
  - Investigational Site Number 840064, New York, New York
  - Investigational Site Number 840005, New York, New York
  - Investigational Site Number 840071, Schenectady, New York
  - Investigational Site Number 840091, Staten Island, New York
  - Investigational Site Number 840045, Syracuse, New York
  - Investigational Site Number 840084, Asheville, North Carolina
  - Investigational Site Number 840078, Charlotte, North Carolina
  - Investigational Site Number 840042, Raliegh, North Carolina
  - Investigational Site Number 840105, Sanford, North Carolina
  - Investigational Site Number 840074, Wilmington, North Carolina
  - Investigational Site Number 840090, Winston-Salem, North Carolina
  - Investigational Site Number 840041, Bismarck, North Dakota
  - Investigational Site Number 840003, Canton, Ohio
  - Investigational Site Number 840009, Dayton, Ohio
  - Investigational Site Number 840053, Monaca, Pennsylvania
  - Investigational Site Number 840056, Philadelphia, Pennsylvania
  - Investigational Site Number 840072, Cranston, Rhode Island
  - Investigational Site Number 840048, Nashville, Tennessee
  - Investigational Site Number 840035, Tullahoma, Tennessee
  - Investigational Site Number 840060, Dallas, Texas
  - Investigational Site Number 840052, Mansfield, Texas
  - Investigational Site Number 840028, San Antonio, Texas
  - Investigational Site Number 840070, Henrico, Virginia
  - Investigational Site Number 840109, Richmond, Virginia
  - Investigational Site Number 840017, Roanoke, Virginia
  - Investigational Site Number 840054, Vienna, Virginia
  - Investigational Site Number 840069, Spokane, Washington
  - Investigational Site Number 840079, Morgantown, West Virginia
  - Investigational Site Number 840038, Milwaukee, Wisconsin
  - Investigational Site Number 840112, Milwaukee, Wisconsin
  - Investigational Site Number 840076, Neenah, Wisconsin
- Austria (2):
  - Investigational Site Number 040-001, Linz
  - Investigational Site Number 040-002, Vienna
- Belgium (8):
  - Investigational Site Number 056006, Brasschaat
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056003, Edegem
  - Investigational Site Number 056002, Kortrijk
  - Investigational Site Number 056007, Leuven
  - Investigational Site Number 056008, Liège
  - Investigational Site Number 056009, Liège
  - Investigational Site Number 056005, Melsbroek
- Canada (2):
  - Investigational Site Number 124006, Cambridge
  - Investigational Site Number 124007, St. John's
- Chile (3):
  - Investigational Site Number 152003, Concepción
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152005, Santiago
- Finland (5):
  - Investigational Site Number 246004, Hämeenlinna
  - Investigational Site Number 246005, Kuopio
  - Investigational Site Number 246006, Oulu
  - Investigational Site Number 246001, Turku
  - Investigational Site Number 246003, Turku
- France (37):
  - Investigational Site Number 250002, Agen
  - Investigational Site Number 250003, Aix-en-Provence
  - Investigational Site Number 250004, Albi
  - Investigational Site Number 250005, Amiens
  - Investigational Site Number 250006, Bayonne
  - Investigational Site Number 250007, Bordeaux
  - Investigational Site Number 250008, Caen
  - Investigational Site Number 250009, Cahors
  - Investigational Site Number 250011, Chambéry
  - Investigational Site Number 250012, Colmar
  - Investigational Site Number 250001, Dijon
  - Investigational Site Number 250015, Grenoble
  - Investigational Site Number 250017, Le Mans
  - Investigational Site Number 250018, Lille
  - Investigational Site Number 250019, Limoges
  - Investigational Site Number 250020, Lyon
  - Investigational Site Number 250021, Marseille
  - Investigational Site Number 250022, Metz-Tessy
  - Investigational Site Number 250023, Montbéliard
  - Investigational Site Number 250024, Montpellier
  - Investigational Site Number 250025, Mulhouse
  - Investigational Site Number 250026, Nancy
  - Investigational Site Number 250027, Nantes
  - Investigational Site Number 250028, Nîmes
  - Investigational Site Number 250016, Paris
  - Investigational Site Number 250029, Paris
  - Investigational Site Number 250043, Pau
  - Investigational Site Number 250031, Quimper
  - Investigational Site Number 250032, Reims
  - Investigational Site Number 250033, Rouen
  - Investigational Site Number 250030, Saint-Germain-en-Laye
  - Investigational Site Number 250035, Strasbourg
  - Investigational Site Number 250037, Toulouse
  - Investigational Site Number 250038, Tours
  - Investigational Site Number 250039, Valence
  - Investigational Site Number 250040, Valenciennes
  - Investigational Site Number 250013, Vichy
- Germany (3):
  - Investigational Site Number 276001, Bergisch Gladbach
  - Investigational Site Number 276003, Berlin
  - Investigational Site Number 276004, Freiburg im Breisgau
- Greece (4):
  - Investigational Site Number 300002, Athens
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300005, Larissa
  - Investigational Site Number 300004, Thessaloniki
- Italy (7):
  - Investigational Site Number 380008, Ancona
  - Investigational Site Number 380009, Bari
  - Investigational Site Number 380002, Gallarate (VA)
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380004, Milan
  - Investigational Site Number 380006, Napoli
  - Investigational Site Number 380005, Orbassano (TO)
- Norway (3):
  - Investigational Site Number 578002, Bergen
  - Investigational Site Number 578003, Namsos
  - Investigational Site Number 578001, Oslo
- Spain (8):
  - Investigational Site Number 724004, A Coruña
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724010, Córdoba
  - Investigational Site Number 724008, Donostia / San Sebastian
  - Investigational Site Number 724001, El Palmar (murcia)
  - Investigational Site Number 724006, Santiago de Compostela
  - Investigational Site Number 724007, Valencia
  - Investigational Site Number 724005, Valladolid
- Sweden (3):
  - Investigational Site Number 752001, Karlstad
  - Investigational Site Number 752003, Kungsbacka
  - Investigational Site Number 752002, Motala
- United Kingdom (9):
  - Investigational Site Number 826-005, Birmingham
  - Investigational Site Number 826-003, Brighton
  - Investigational Site Number 826-007, Glasgow
  - Investigational Site Number 826-008, Leeds
  - Investigational Site Number 826-010, Leicester
  - Investigational Site Number 826-009, London
  - Investigational Site Number 826-001, Norwich
  - Investigational Site Number 826-006, Romford
  - Investigational Site Number 826-004, Salford

REFERENCES:
- [Derived] Coyle PK, Khatri B, Edwards KR, Meca-Lallana JE, Cavalier S, Rufi P, Benamor M, Poole EM, Robinson M, Gold R. Teriflunomide real-world evidence: Global differences in the phase 4 Teri-PRO study. Mult Scler Relat Disord. 2019 Jun;31:157-164. doi: 10.1016/j.msard.2019.03.022. Epub 2019 Mar 30. PMID 31005729
- [Derived] Coyle PK, Khatri B, Edwards KR, Meca-Lallana JE, Cavalier S, Rufi P, Benamor M, Brette S, Robinson M, Gold R; Teri-PRO Trial Group. Patient-reported outcomes in relapsing forms of MS: Real-world, global treatment experience with teriflunomide from the Teri-PRO study. Mult Scler Relat Disord. 2017 Oct;17:107-115. doi: 10.1016/j.msard.2017.07.006. Epub 2017 Jul 6. PMID 29055438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 169 centers in 14 countries. A total of 1102 participants were screened between June 14, 2013 and November 27, 2014 of whom 101 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: A total of 1001 participants were included and 1000 participants were treated in the study. Dose of Teriflunomide tablet was given according to local labelling 14 mg or 7 mg (Teriflunomide 14 mg was the recommended dosage worldwide, except in the US [where both 7 mg and 14 mg were available]).
Period: Overall Study
Arm/Group | Teriflunomide
Started | 1001
Treated | 1000
Completed | 786
Not Completed | 215
Not completed — Adverse Event | 106
Not completed — Lack of Efficacy | 53
Not completed — Poor Compliance to Protocol | 11
Not completed — Included But Not treated | 1
Not completed — Other than Specified Above | 44

BASELINE CHARACTERISTICS:
Population: Baseline population included all treated participants.
Groups:
- Teriflunomide: Teriflunomide 14 mg or 7 mg according to local labelling QD orally for 48 weeks.
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 756
  Male | 244

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Version 1.4 - Assessment of Global Satisfaction Subscale Score With Teriflunomide Treatment at Week 48
Description: TSQM version 1.4 is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. It comprises of 14 items assessing the following 4 domains: effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions:12-14).
  Primary outcome was the global satisfaction score. The score of the corresponding item was added based on the algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain.
Time Frame: Week 48
Population: Efficacy population that included all treated participants. Number of participants analyzed = participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 889
units on a scale | 68.17 (27.66)

2. Secondary Outcome: Change From Baseline in TSQM Scores in Participants Switching From Another Disease Modifying Therapy (DMT) at Week 4 and Week 48
Description: TSQM version 1.4 is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. It comprises of 14 items assessing the following 4 domains: effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions: 12-14). For each of the 4 domains the scores of the corresponding items were added based on an algorithm to create a score of 0 to 100. Higher scores indicated greater satisfaction .
Time Frame: Baseline, Week 4, Week 48
Population: Analysis was performed on Efficacy population. Number of participants analyzed=participants with available data at specified time point. Here, 'n' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 594
units on a scale
  Global Satisfaction Score Change at Week 4 (n=482) | 21.35 (27.51)
  Global Satisfaction Score Change at Week 48(n=457) | 16.55 (34.29)
  Effectiveness Score Change at Week 4 (n=477) | 12.02 (25.53)
  Effectiveness Score Change at Week 48 (n=453) | 10.19 (28.90)
  Side effects Score Change at Week 4 (n=479) | 24.31 (35.47)
  Side effects Score Change at Week 48 (n=456) | 19.95 (39.00)
  Convenience Score Change at Week 4 (n=487) | 34.64 (26.37)
  Convenience Score Change at Week 48 (n=461) | 32.21 (27.01)

3. Secondary Outcome: Change From Week 4 in TSQM Scores in Naïve Participants to Week 48
Description: TSQM version 1.4 is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. It comprises of 14 items assessing the following 4 domains: effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions: 12-14). For each of the 4 domains the scores of the corresponding items were added based on an algorithm to create a score of 0 to 100. Higher scores indicated greater satisfaction.
Time Frame: Week 4, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 285
units on a scale
  Change in Global Satisfaction Score (n=234) | -1.34 (23.59)
  Change in Effectiveness Score (n=231) | 1.76 (27.48)
  Change in Side effects Score (n=234) | -5.44 (25.11)
  Change in Convenience Score (n=235) | 0.33 (12.96)

4. Secondary Outcome: Change From Baseline in Disease Progression Using Patient Determined Disease Steps (PDDS) Score at Week 48
Description: PDDS scale developed to assess the disability in Multiple Sclerosis (MS) participants and in assessing disease progression that focuses mainly on how participants walk. PDDS scale consists of 0 = normal; 1 = mild disability; 2 = moderate disability; 3 = gait disability; 4 = early cane; 5 = late cane; 6 = bilateral support; 7 = wheelchair/scooter and 8 = bedridden. A higher score represented higher level of disability.
Time Frame: Baseline, Week 48
Population: Analysis was performed on Efficacy population. Number of participants analyzed=participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 860
units on a scale | -0.01 (1.05)

5. Secondary Outcome: Change From Baseline in Multiple Sclerosis Performance Scale (MSPS) Score at Week 24 and Week 48
Description: MSPS was a self-reported measure for MS associated disability in which participants were asked to indicate the category that best described their condition during the past month on the following 8 subscales: mobility, hand function, vision, fatigue, cognitive symptoms, bladder/bowel, sensory symptoms and spasticity symptoms. MSPS used a single question to assess each of 8 subscales. All of the subscales ranged from 0= normal to 5= total disability, except mobility subscale which ranged from 0= normal to 6=total disability. Total MSPS score ranged from 0 =normal to 41=greater disability, where higher score reflected greater disability.
Time Frame: Baseline, Week 24, Week 48
Population: Analysis was performed on Efficacy population. Here, 'n' signifies number of participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
units on a scale
  Change at Week 24 (n=854) | -0.61 (3.89)
  Change at Week 48 (n=875) | -0.06 (4.33)

6. Secondary Outcome: Annualized Treated Relapse Rate
Description: Annualized treated relapse rate was defined as the total number of treated relapses during the study treatment period divided by the total number participants-years of treatment. Only events occurred during the treatment period (first drug administration to last drug administration) were considered for analysis.
Time Frame: Baseline up to end of treatment (up to Week 48)
Population: Analysis was performed on Efficacy population.
Measure: Number; unit: relapses per patient-year
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
relapses per patient-year | 0.200

7. Secondary Outcome: Time to Relapse: Kaplan-Meier Estimates of the Probability of Treated Relapse at Week 4, Week 24 and Week 48
Description: A treated relapse was defined as a relapse treated by a systemic corticosteroid treatment or by another DMT. If a participant had no treated relapse before treatment discontinuation/completion, then the participant was considered as free of treated relapse until the date of treatment discontinuation/completion. Only treated relapse occurred during the treatment period (first drug administration to last drug administration) were considered for analysis. Kaplan-Meier method was used to estimate the probability of treated MS relapse at 4, 24 and 48 weeks.
Time Frame: Baseline up to end of treatment (up to Week 48)
Population: Analysis was performed on Efficacy population.
Measure: Number (95% Confidence Interval); unit: percent probability of treated relapse
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
percent probability of treated relapse
  Percent Probability of Treated Relapse at Week 4 | 1.8 [1.0 to 2.6]
  Percent Probability of Treated Relapse at Week 24 | 9.4 [7.5 to 11.2]
  Percent Probability of Treated Relapse at Week 48 | 15.5 [13.2 to 17.9]

8. Secondary Outcome: Change From Baseline in Cognition Measured by Symbol Digit Modalities Test (SDMT) Score at Week 48
Description: SDMT measures the time to pair abstract symbols with specific numbers. It is a simple substitution task that gives the examinee 90 seconds to pair specific numbers with given geometric figures as a measure for screening cognitive impairment. The score is computed as a ratio of number of correct responses divided by the total number of responses. The test score range from 0 (worst outcome) to 1 (best outcome). Higher scores are indicative of better cognition function.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 854
units on a scale | 0.00 (0.06)

9. Secondary Outcome: Overview of Adverse Events (AEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during from first study drug intake up to 112 days after last intake for participant with no accelerated elimination procedure (AEP) or to last AEP follow up visit for participants with AEP. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: From first study drug intake up to 112 days after last intake for participant with no AEP or to last AEP follow up visit for participants with AEP
Population: Safety Population that included all treated participants who received at least 1 dose or part of a dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
percentage of participants
  Any TEAE | 82.3
  Any treatment emergent SAE | 12.7
  Any TEAE leading to death | 0.4
  Any TEAE leading to permanent discontinuation | 10.9

10. Secondary Outcome: Percentage of Participants With Treatment Compliance of ≥80% During the Study Treatment Period
Description: Percentage of compliance for a participant was defined as the number of days that the participant was compliant (1 tablet/day) divided by the exposure duration in days (from the first dose administration to the last dose administration) times 100.
Time Frame: Baseline up to end of treatment (up to Week 48)
Population: Analysis was performed on Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
percentage of participants | 98.2

11. Secondary Outcome: Duration of Teriflunomide Treatment Exposure
Description: Duration of exposure was defined as last dose date - first dose date + 1 day, regardless of unplanned intermittent discontinuations and regardless of dosage administered (14 mg or 7 mg).
Time Frame: Baseline up to end of treatment (up to Week 48)
Population: Analysis was performed on Safety population.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
Days | 301.6 (89.1)

12. Secondary Outcome: Change From Baseline in Multiple Sclerosis International Quality of Life (MusiQoL) Score at Week 48
Description: The MusiQoL is a quality of life questionnaire that consists of 31 questions, divided into 9 dimensions: activities of daily living, physiological well-being, symptoms, relationship with friends, relationship with family, sentimental and sexual life, coping, rejection and relationship with healthcare system. All the 9 dimension scores and the global scores are linearly transformed and standardized on 0 (worst outcome) -100 (best outcome) scale. Higher scores represents higher quality of life.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 826
units on a scale | 0.99 (10.82)

13. Secondary Outcome: Change From Baseline in Stern Leisure Activity Scale at Week 48
Description: The Stern Leisure Activity Scale is a self-reported scale that consists of 13 questions assessing the participant's participation in leisure activities during the preceding month. One point is given for participation in each of the 13 activities and an aggregate score (range from 0 to 13) is obtained. ≤ 6 score is considered as low leisure activity and > 6 score as high leisure activity.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 845
units on a scale | 0.07 (1.93)

14. Secondary Outcome: Expanded Disability Status Scale (EDSS) Score at Baseline and Week 48
Description: EDSS is a method of quantifying disability in MS participants and monitoring changes in the level of disability over time. EDSS quantifies disability in 8 functional systems: pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other. EDSS scale ranges from 0 to 10 in 0.5 unit increments that represents higher levels of disability. EDSS score 1.0 to 4.5 refers to people with MS who are fully ambulatory; EDSS score 5.0 to 9.5 refers to impairment to ambulation; EDSS score 10 refers to death due to MS.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriflunomide
Number analyzed (Participants) | 1000
units on a scale
  Baseline (n=981) | 3.05 (1.94)
  Week 48 (n=886) | 3.05 (1.98)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to the last visit (Week 52) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are TEAEs that is AEs that developed/worsened from first study drug intake up to 112 days after last intake for participant with no AEP or to last AEP follow up visit for participants in AEP. Analysis was performed on safety population.
Arm/Group | Teriflunomide
Serious Adverse Events (participants affected / at risk) | 127/1000
Other Adverse Events (participants affected / at risk) | 498/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teriflunomide (N=1000)
Neutropenia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blindness Unilateral (Eye disorders) | 1
Retinal Artery Thrombosis (Eye disorders) | 1
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1
Colitis Microscopic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2
Hiatus Hernia (Gastrointestinal disorders) | 2
Volvulus (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 3
Non-Cardiac Chest Pain (General disorders) | 3
Oedema Peripheral (General disorders) | 1
Bile Duct Stone (Hepatobiliary disorders) | 1
Biliary Colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium Difficile Colitis (Infections and infestations) | 1
Clostridium Difficile Infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Myelitis (Infections and infestations) | 1
Oesophageal Candidiasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pelvic Abscess (Infections and infestations) | 1
Perichondritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Viral Infection (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 6
Blood Pressure Increased (Investigations) | 1
Clostridium Test Positive (Investigations) | 1
Fibrin D Dimer Increased (Investigations) | 1
Transaminases Increased (Investigations) | 1
Weight Decreased (Investigations) | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Small Cell Lung Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Carpal Tunnel Syndrome (Nervous system disorders) | 1
Cerebral Sarcoidosis (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Cervicobrachial Syndrome (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Medication Overuse Headache (Nervous system disorders) | 1
Multiple Sclerosis (Nervous system disorders) | 2
Multiple Sclerosis Relapse (Nervous system disorders) | 21
Neuromyelitis Optica (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Toxic Encephalopathy (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Trigeminal Neuralgia (Nervous system disorders) | 2
Uhthoff's Phenomenon (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Acute Psychosis (Psychiatric disorders) | 1
Adjustment Disorder With Depressed Mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Suicidal Ideation (Psychiatric disorders) | 1
Suicide Attempt (Psychiatric disorders) | 2
Acute Kidney Injury (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Hypertonic Bladder (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 2
Acute Interstitial Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung Cyst (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Abdominoplasty (Surgical and medical procedures) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Essential Hypertension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teriflunomide (N=1000)
Diarrhoea (Gastrointestinal disorders) | 172
Nausea (Gastrointestinal disorders) | 82
Fatigue (General disorders) | 52
Nasopharyngitis (Infections and infestations) | 54
Urinary Tract Infection (Infections and infestations) | 62
Alanine Aminotransferase Increased (Investigations) | 57
Headache (Nervous system disorders) | 68
Alopecia (Skin and subcutaneous tissue disorders) | 229

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.